CLINICAL TRIAL: NCT01437254
Title: A Phase I Study of Cyclotron-produced Tc-99m Pertechnetate (CPERT) in Patients With Thyroid Cancer
Brief Title: To Compare Safety and the General Imaging Pattern of Cyclotron Produced Technetium vs. Generator Produced Technetium in Patients With Thyroid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Natural Resources, Canada (Unknown); Edmonton PET Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DX-CPERT-001
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Thyroid Neoplasms
Keywords: 99mTc Pertechnetate; thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Nuclear Medicine physicians interpreting the whole body biodistribution pattern of CPERT and GPERT scans were blinded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm Number 1 CPERT (Experimental): 1 CPERT scan, blood and vital sign collection
  Interventions: Drug: CPERT
- Arm Number 2 GPERT (Active Comparator): 1 GPERT Scan
  Interventions: Drug: GPERT

INTERVENTIONS:
Drug: CPERT — Single 340 MBq CPERT scan in first 10 subjects
  Arms: Arm Number 1 CPERT
Drug: GPERT — Single 340 MBq GPERT scan in up to 20 case-matched controls
  Arms: Arm Number 2 GPERT

SUMMARY:
The cyclotron production model of Tc-99m pertechnetate (CPERT) has received significant validation in the independent expert review conducted by Natural Resources Canada (NRCan) in the follow up to the Chalk River crisis. The University of Alberta's Edmonton PET Centre and the Edmonton Radiopharmaceutical Centre is a cyclotron / radiopharmacy unit, providing a safe, cost effective, unsubsidized, and reliable supply of radiopharmaceuticals to hospitals and clinics in Edmonton and northern Alberta. A Phase I study is proposed to show safety of CPERT as well as comparability with generator-produced Tc-99m pertechnetate (GPERT) in subjects with well differentiated thyroid carcinoma post-thyroidectomy and prior to planned I-131 Iodide treatment.

DETAILED DESCRIPTION:
Patients who have had a thyroidectomy for cancer routinely have a Tc-99m Pertechnetate (GPERT) scan at the Cross Cancer Institute to check for thyroid tissue remnants prior to radioactive iodine therapy. The first 10 subjects will receive a CPERT whole body scan, and and 20 subsequent case-matched controls (2 for each CPERT subject, matched for age and gender) will receive a GPERT whole body scan. CPERT safety will be assessed by pre-injection and post-imaging collection of vital signs and blood samples (haematology and biochemistry). Adverse event collection will be done for both CPERT and GPERT subjects. The whole body biodistribution pattern of CPERT will be qualitatively compared to GPERT by two independent and blinded Nuclear Medicine physicians.

ELIGIBILITY:
Inclusion Criteria:

* If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test is required.
* Have confirmed well differentiated thyroid cancer, post-thyroidectomy and pre-RAI
* Biochemical parameters as measured are required to be within 5 times the normal limits for age
* white blood cell count (WCB) > 3.0/µL
* absolute neutrophil count (ANC) > 1.5/µL
* Platelets > 75,000/µL
* Hemoglobin > 10 g/dL
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in the study
* Karnofsky Performance Scale score of 50 - 100

Exclusion Criteria:

* Nursing or pregnant females
* Biochemical parameters as measured outside 5 times the normal limits for age within 14 days of the pre-treatment scan
* White blood cell count (WCB < 3.0/µL)
* absolute neutrophil count (ANC) < 1.5/µL
* Platelets < 75,000/µL
* Haemoglobin < 10 g/dL
* unable and unwilling to follow instructions and comply with the protocol
* unable or unwilling to provide written informed consent prior to participation in the study
* Karnofsky Performance Scale score <50

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety of CPERT | 7 months
  CPERT safety will be assessed by evaluation of vital signs (pre-injection and post-imaging), blood haematology (pre-injection and post-imaging), SMA-12 clinical biochemistry profile (pre-injection and post-imaging) and collection of adverse events.

SECONDARY OUTCOMES:
Comparison of general biodistribution of CPERT and GPERT. | 7 months
  The whole body biodistribution pattern of CPERT will be compared to GPERT using two independent and blinded Nuclear Medicine physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MB, FCRPC, Principal Investigator — Professor, Department of Oncology
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada